CLINICAL TRIAL: NCT03856905
Title: Extracorporeal Shock Wave Therapy Versus Functional Electrical Stimulation on Spasticity, Function and Gait Parameters in Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mahmoud Eid, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NU/MID/16/025
Record Dates: First submitted 2019-02-23; First posted 2019-02-27 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Children With Cerebral Palsy
Keywords: Cerebral palsy; Extracorporeal Shock Wave Therapy; Functional Electrical Stimulation; Function; Gait; Spasticity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical therapy group (Active Comparator): The children in this group will receive the conventional physical therapy program (CPTP). It will consist of gentle stretching exercises for spastic muscles, facilitation of muscle contraction for the anti-spastic muscles, proprioceptive training, balance and postural control exercises, neuro-developmental techniques, and gait training. The total program will be conducted for 1 h, three sessions/week for 12 weeks.
  Interventions: Other: Physical therapy program
- Extra-corporeal shock wave therapy group (Experimental): The children in this group only will receive the extra-corporeal shock wave therapy (ESWT). An electromagnetic coil lithotripter (Modulith SLK; Storz Medical AG, Tagerwillen, Switzerland) provided with in-line ultrasound, radiographic, and computerized aiming (Lithotrack system; Storz Medical AG) will be used. The energy applied will be 0.030 mJ/mm2. The frequency will be 5 Hz, with a pressure of 1.5 bars, burst mode, one session/week for 12 weeks. The treatment is painless and does not require any kind of anesthesia or the use of analgesic drugs
  Interventions: Other: Physical therapy program; Device: Extracorporeal shock wave therapy
- Functional electrical stimulation group (Experimental): The children in this group will receive the functional electrical stimulation (FES). The FES will be applied by using the WalkAide system (Innovative Neurotronics, Austin, TX, USA).
  The stimulation parameters will include pulse frequency (16-33 pulses per second), pulse width (25-300 µs) to produce a desired movement as close to normal as possible at the ankle during gait.
  Interventions: Other: Physical therapy program; Device: Functional electrical stimulation

INTERVENTIONS:
Other: Physical therapy program — It will consist of gentle stretching exercises for spastic muscles, facilitation of muscle contraction for the anti-spastic muscles, proprioceptive training, balance and postural control exercises, neurodevelopmental techniques, and gait training.
Device: Extracorporeal shock wave therapy — It is an electromagnetic coil lithotripter (Modulith SLK; Storz Medical AG, Tagerwillen, Switzerland) provided with in-line ultrasound, radiographic, and computerized aiming (Lithotrack system; Storz Medical AG). The energy applied will be 0.030 mJ/mm2. The frequency will be 5 Hz, with a pressure of 1.5 bars, burst mode.
  Arms: Extra-corporeal shock wave therapy group
Device: Functional electrical stimulation — It is a highly advanced medical device that consists of a battery-operated, single-channel electrical stimulator, two electrodes, and electrode leads with a cuff holds the system in place. The stimulation parameters will include pulse frequency (16-33 pulses per second), pulse width (25-300 µs) to produce a desired movement as close to normal as possible at the ankle during gait.
  Arms: Functional electrical stimulation group

SUMMARY:
Objective: The purpose of this study will compare the effects of extracorporeal shock wave therapy (ESWT) versus functional electrical stimulation (FES) on spasticity, function and gait parameters in hemiplegic cerebral palsy (CP).

Methods: Forty-five children with CP ranging in age from 6 to 9 years will be selected and will participate in this study. They will be assigned randomly using opaque envelopes into three groups (A, B and C). Group A will consist of 15 children and will receive the conventional physical therapy program (CPTP) in addition to ankle foot orthosis (AFO). Group B will consist of 15 children and will receive the CPTP, AFO in addition to ESWT. Group C also will consist of 15 children and will receive the CPTP, AFO in addition to FES. The program of treatment will be 3 days/week for 12 weeks. Assessment of spasticity by using the modified ashworth scale (MAS), function by using the pediatric functional independence scale and gait parameters by using the 3-dimensional gait analysis will be conducted at baseline and after 12 weeks of the treatment program.

DETAILED DESCRIPTION:
Forty-five children with cerebral palsy (CP) with ages ranging from 6 to 9 years will participate in this study. They will be selected from the out-patient clinic of Obstetric and Pediatric Hospital, Comprehensive Rehabilitation Center, King Khalid Hospital and Najran Generalized Hospital, Najran, KSA, according to inclusive criteria including, children who demonstrate unilateral dynamic equinus deformity, all children must be ambulant independently and they will classified at Gross Motor Function Classification System (GMFCS) levels I or II. They must be free from any skeletal abnormalities other than spasticity and the degree of spasticity according to the Modified Ashworth Scale (MAS) within the range of 1+ and 2 grades. Moreover, all children must have a minimum five degrees of passive ankle dorsiflexion with knee joint extended. Exclusion criteria including, the use of botulinum toxin injection of the planter flexor muscles within the 4 months before the study and orthopedic surgery to the ankle joint in the previous 6 months before or during the study.

Children will be assigned randomly using opaque envelopes into three intervention groups (A, B and C). Group A will receive the conventional physical therapy program (CPTP) in addition to ankle foot orthosis (AFO). Group B will receive the CPTP, AFO in addition to Extra-corporeal shock wave therapy (ESWT), whereas group C will receive CPTP, AFO in addition to functional electrical stimulation (FES). All groups will receive the treatment program 3 sessions/week for 12 weeks. Evaluation of spasticity by using the MAS, function by using the pediatric functional independence scale and gait parameters by using the 3-dimensional gait analysis will be conducted before and after 12 weeks of the treatment program.

ELIGIBILITY:
Inclusion Criteria:

* children who demonstrate unilateral dynamic equinus deformity,
* All children must be ambulant independently and they will classified at Gross Motor Function Classification System (GMFCS) levels I or II,
* They must be free from any skeletal abnormalities other than spasticity and the degree of spasticity according to the Modified Ashworth Scale (MAS) within the range of 1+ and 2 grades,
* Moreover, all children must have a minimum five degrees of passive ankle dorsiflexion with knee joint extended

Exclusion Criteria:

* The use of botulinum toxin injection of the planter flexor muscles within the 4 months before the study,
* Orthopedic surgery to the ankle joint in the previous 6 months before or during the study.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Spasticity (assessing change between baseline and after treatment) | This outcome will be measured for each child before the beginning of treatment program and immediately after 12 weeks of the treatment program
  Name of the scale: The Modiﬁed Ashworth Scale. It will be used to measure spasticity of the ankle plantar ﬂexors. It is a simple measure of spasticity giving grades (0, 1, 1+, 2, 3, 4) 0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension The total score will be obtained by calculating the mean of the obtained data Lower scores indicate better results.
Function (assessing change between baseline and after treatment) | This outcome will be measured for each child before the beginning of treatment program and immediately after 12 weeks of the treatment program.
  Name of the scale: Functional Independence Measure for Children It will be used to assess the functions of children between 6 months and 12 years.
  The scores of the scale extends from minimum 18 (fully dependent) to maximum 126 (fully independent) The scale measures different functional activities in children and the total score will be obtained for each category by computing the mean of the obtained data.
  Higher scores indicate better results.
Cadence (assessing change between baseline and after treatment) | This outcome will be measured for each child before the beginning of treatment program and immediately after 12 weeks of the treatment program.
  Cadence will be evaluated by using the 3-dimensional motion analysis system (Qualisys; Qualisys Inc, Goeteborg, Sweden).
  The unit of measure of cadence: steps/minute
Stride length (assessing change between baseline and after treatment) | This outcome will be measured for each child before the beginning of treatment program and immediately after 12 weeks of the treatment program.
  Stride length will be evaluated by using the 3-dimensional motion analysis system (Qualisys; Qualisys Inc, Goeteborg, Sweden).
  The unit of measure of Stride length: meter
Velocity (assessing change between baseline and after treatment) | This outcome will be measured for each child before the beginning of treatment program and immediately after 12 weeks of the treatment program.
  Velocity will be evaluated by using the 3-dimensional motion analysis system (Qualisys; Qualisys Inc, Goeteborg, Sweden).
  The unit of measure of velocity: meter/sec
Ankle dorsiflexion angle (assessing change between baseline and after treatment) | This outcome will be measured for each child before the beginning of treatment program and immediately after 12 weeks of the treatment program.
  Ankle dorsiflexion angle will be evaluated by using the 3-dimensional motion analysis system (Qualisys; Qualisys Inc, Goeteborg, Sweden).
  The unit of measure of Ankle dorsiflexion angle: degrees

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy - Cairo University, Giza, Egypt